CLINICAL TRIAL: NCT04743596
Title: High-definition Videobronchoscopy With Optical Enhancement for the Diagnosis of Endobronchial Sarcoidosis: a Pilot Study
Brief Title: High-definition Videobronchoscopy in Sarcoidosis
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3871
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-02

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sarcoidosis group: Consecutive patients with clinical and radiological (CT scan) suspect of sarcoidosis as assessed by a respiratory physician.
  Interventions: Device: High-Definition Videobronchoscopy

INTERVENTIONS:
Device: High-Definition Videobronchoscopy — Endoscopic inspection and endobronchial biopsy with standard forceps during high-definition videobronchoscopy.

SUMMARY:
In the last few years, high-definition (HD) videobronchoscopy has become widely available in the market and will progressively become the standard of care for airway inspection and sampling, as it provides substantially higher resolution images as compared to conventional white light bronchoscopy. Furthermore, in combination with improved video processor units, some HD videobronchoscopes offer post-processing real-time image enhancement (i-scan technology). Preliminary studies, performed in the setting of lung cancer, suggest that HD bronchoscopy with optical image enhancement (OE) may result in better detection of subtle vascular abnormalities in the airways, which are often associated with preneoplastic lesions. We hypothesize that HD videobronchoscopy could help identify bronchial involvement from sarcoidosis before it is (plainly) visible by conventional bronchoscopy.

DETAILED DESCRIPTION:
Sarcoidosis is a systemic disorder of unknown cause that primarily involves the lung and lymphatic systems and that can be more reliably diagnosed if a compatible clinical picture is combined with a pathologic demonstration of non-necrotizing epithelioid-cell granulomas. As the thorax (bronchi, lung parenchyma, and/or intrathoracic lymph nodes) is almost invariably involved, bronchoscopy with its ancillary sampling procedures (endobronchial biopsy, transbronchial lung biopsy, bronchoalveolar lavage, conventional and ultrasound guided-transbronchial needle aspiration, endoscopic ultrasound with fine needle aspiration) has been the diagnostic tool most frequently used to confirm pathologically the clinical suspect of sarcoidosis.

Among the possible bronchoscopic sampling procedures, endobronchial biopsy (EBB), which is the easiest and safest, has long been used, even though its value has been assessed in small studies, mostly retrospective. Although its diagnostic yield has been shown to be widely variable (5%-71%) across different studies, EBB has constantly demonstrated to increase the diagnostic success of bronchoscopy in sarcoidosis when coupled with other sampling methods. In the last few years, high-definition (HD) videobronchoscopy has become widely available in the market and will progressively become the standard of care for airway inspection and sampling, as it provides substantially higher resolution images as compared to conventional white light bronchoscopy. Furthermore, in combination with improved video processor units, some HD videobronchoscopes offer post-processing real-time image enhancement (i-scan technology). Preliminary studies, performed in the setting of lung cancer, suggest that HD bronchoscopy with optical image enhancement (OE) may result in better detection of subtle vascular abnormalities in the airways, which are often associated with preneoplastic lesions. We hypothesize that HD videobronchoscopy could help identify bronchial involvement from sarcoidosis before it is (plainly) visible by conventional bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. indication to a pathological confirmation of the clinical and radiological (CT) suspect of sarcoidosis;
2. age > 18 years;
3. ASA score 1-3.

Exclusion Criteria:

1. inability to consent;
2. steroid therapy (at least 1 week) in the 2 months preceding bronchoscopy;
3. pregnancy;
4. uncontrolled coagulopathy;
5. contraindication to temporary interruption of anticoagulants or antiplatelet drugs, except aspirin;

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with clinical and radiological (CT scan) suspect of sarcoidosis as assessed by a respiratory physician
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of endobronchial biopsy guided by HD videobronchoscopy for the detection of granulomas | 1 month
  The diagnostic yield will be calculated on a per patient basis (number of patients in whom the pathological examination of endobronchial biopsies shows non necrotizing granulomas/all the patients submitted to endobronchial biopsies)

SECONDARY OUTCOMES:
Prevalence of airway abnormalities in patients with suspected sarcoidosis at HD bronchoscopy | 1 day
  The prevalence of airway abnormalities will be calculated on a per patient basis (number of patients in whom the HD videobronchoscopy shows abnormalities in the endoscopically visible airways/all the patients submitted to HD videobronchoscopy)
Prevalence of different patterns of airway abnormalities in patients with suspected sarcoidosis at HD videobronchoscopy | 1 day
  The following patterns of airway abnormalities, well described in the literature in the setting of endobronchial sarcoidosis, will be evaluated for the assessment of the present endpoint: a) cobblestoning (diffuse, coalescing nodules); b) nodularity (sparse, discrete nodules); c) thickening; d) plaque (infiltrative, raised, flat, white or yellowish areas); e) marked hyperaemia. In those cases in which airway abnormalities are detected, but they do not fall into any of the above patterns, they will be classified into a 6th pattern named "miscellanea".
Specificity for the detection of granulomas of the above 6 different patterns of airway abnormalities identified during HD bronchoscopy | 1 month
  This endpoint will be calculated on a per-lesions basis (number of cases of airway abnormality referring to one the 6 predefined patterns in which the pathological examination of endobronchial biopsies shows non necrotizing granulomas/all the airway abnormalities referring to that specific predefined pattern submitted to endobronchial biopsy).
The interobserver agreement for the identification of the above 6 predefined patterns of airway abnormalities. | 1 month
  At the end of the study, the videos referring to each endobronchial abnormality submitted to biopsy in each enrolling center will be independently classified by two interventional pulmonologist blinded to the clinical, radiological and pathological findings.
Diagnostic yield for the detection of endobronchial granulomas according to clinical, radiological and endoscopic findings. | 6 months
  The association between the following findings and the diagnostic yield of EBBs will be assessed: sex; ethnicity; sarcoidosis stage (I-IV); presence versus absence of endobronchial abnormalities at HD bronchoscopy; pattern of airway abnormality at HD bronchoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Trisolini, MD, Principal Investigator — Catholic University of the Sacred Hearth
Locations (5):
- Italy (2):
  - Azienda Ospedaliero Universitaria di Bologna, Bologna
  - Fondazione Policlinico Univeristario A. Gemelli IRCCS, Roma
- Academic Medical Centre, Amsterdam, Netherlands
- Russia (2):
  - Central TB Research Institute, Moscow
  - Research Institute of TB and Thoracic Surgery, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Livi V, Sivokozov I, Annema JT, Candoli P, Vasilev I, Kramer T, Ferrari M, Madan K, Fielding D, Murgu S, Cancellieri A, Semyonova LA, Puci M, Sotgiu G, Trisolini R. High-Definition Videobronchoscopy for the Diagnosis of Airway Involvement in Sarcoidosis: The Enhance Sarcoidosis Multicenter Study. Chest. 2023 Nov;164(5):1243-1252. doi: 10.1016/j.chest.2023.04.034. Epub 2023 Apr 28. PMID 37121391